CLINICAL TRIAL: NCT05496114
Title: The Impact of Medical Checklists on the Management of Acute Situations in the Emergency Department. A Simulation-based Randomised Controlled Trial.
Brief Title: Medical Checklists in the Emergency Department
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Malu van der Capellen, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: W22_163
Record Dates: First submitted 2022-08-08; First posted 2022-08-11 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Emergencies; Tricyclic Antidepressant Poisoning; Tricyclic Antidepressant Toxicity
Keywords: Medical checklists
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Intervention Model Description: Participants (emergency physicians) will be allocated to performing the scenario with or without checklist in a randomized fashion on a 1:1 ratio. Computerized randomization will take place using an online randomization module.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group: with checklist (Experimental): When starting the scenario, a checklist will be given to the emergency physician. The checklist outlines interventions to consider during management of a patient with tricyclic antidepressant poisoning. Each checklist will include indications, contra-indications and for medication, dose, route and rate of administration.
  Interventions: Device: Checklist
- Control group: without checklist (No Intervention): Emergency physicians will be asked to perform the scenario as they would in their daily practice. They will be allowed to use their usual cognitive aids (eg, phone, internet) but not allowed to request help from others.

INTERVENTIONS:
Device: Checklist — A checklist is an aid that outlines assessments or actions systematically. In this study, the checklist outlines interventions to consider during management of a patient with tricyclic antidepressant poisoning. Each checklist will include indications, contra-indications and for medication, dose, route and rate of administration.
  Arms: Intervention group: with checklist

SUMMARY:
This study aims to investigate whether the use of medical checklists in the emergency department can decrease resuscitation time in critically ill patients.

DETAILED DESCRIPTION:
A scenario evaluating tricyclic antidepressant poisoning will be carried out with and without medical checklist access. Emergency physicians from the Netherlands who are willing to take part in the study are randomly allocated to perform the scenario with or without checklists.

ELIGIBILITY:
Inclusion Criteria:

* Emergency Physicians recognised by KNMG (Koninklijke Nederlandsche Maatschappij tot bevordering van de Geneeskunst) working in the Netherlands

Exclusion Criteria:

* Residents (in Dutch: AIOS) Emergency Medicine
* Interns (in Dutch: ANIOS) Emergency Medicine

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Duration of the scenario | Through study completion, indicated 10 months
  The primary outcome is the duration of primary resuscitation utilizing the checklists versus treatment on discretion of the treating physician. The simulation will be terminated when all indicated interventions are performed, when the team expresses that they cannot think of any other intervention to perform or when 15 minutes have elapsed.

SECONDARY OUTCOMES:
Number of indicated interventions performed by the emergency physician | Through study completion, indicated 10 months
  Based on the checklist, a number of predefined indicated interventions is established. When reviewing the video recordings, it will be noted whether indicated interventions were performed and when these interventions were performed. The order according to which interventions are performed will not impact on this secondary outcome.
Satisfaction of emergency physicians with the checklists | Through study completion, indicated 10 months
  Participants, who run the scenarios with checklist access, will be asked to fill out a questionnaire evaluating the checklist (5-point Likert scales).

CONTACTS AND LOCATIONS:
Overall Officials: Malu van der Capellen, MD, Principal Investigator — Amsterdam University Medical Center
Locations (1):
- Amsterdam University Medical Center, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dryver E, Lundager Forberg J, Hard Af Segerstad C, Dupont WD, Bergenfelz A, Ekelund U. Medical crisis checklists in the emergency department: a simulation-based multi-institutional randomised controlled trial. BMJ Qual Saf. 2021 Sep;30(9):697-705. doi: 10.1136/bmjqs-2020-012740. Epub 2021 Feb 17. PMID 33597283